CLINICAL TRIAL: NCT02559440
Title: Combination Therapy With Mometasone Furoate and Oxymetazoline in the Treatment of Adenoid Hypertrophy Concomitant With Allergic Rhinitis
Brief Title: Mometasone Furoate and Oxymetazoline in the Treatment of Adenoid Hypertrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Wenlong Liu, Research secretary, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81500772
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Adenoidal Hypertrophy
MeSH Terms: interventions — Mometasone Furoate; Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- mometasone furoate (Active Comparator): In the first treatment stage, 120 children were assigned to mometasone furoate (50μg, 1 puff in each nostril every evening) after two week's run-in period.
  Interventions: Drug: mometasone furoate
- Placebo (Placebo Comparator): In the first treatment stage, 120 children were assigned to control group (normal saline) after two week's run-in period.
  Interventions: Drug: Placebo
- Oxymetazoline + Placebo (Active Comparator): Stage two is a parallel, randomized, double-blind, double-dummy study. Non-responders underwent 2-week washout period and were randomly assigned to groups receiving Oxymetazoline and placebo.
  Interventions: Drug: Oxymetazoline + Placebo
- Placebo + placebo (Placebo Comparator): Stage two is a parallel, randomized, double-blind, double-dummy study. Non-responders underwent 2-week washout period and were randomly assigned to groups receiving placebo and placebo.
  Interventions: Drug: Placebo + placebo
- mometasone furoate + Placebo (Active Comparator): Stage two is a parallel, randomized, double-blind, double-dummy study. Non-responders underwent 2-week washout period and were randomly assigned to groups receiving mometasone furoate and placebo.
  Interventions: Drug: mometasone furoate + Placebo
- mometasone furoate + Oxymetazoline (Active Comparator): Stage two is a parallel, randomized, double-blind, double-dummy study. Non-responders underwent 2-week washout period and were randomly assigned to groups receiving mometasone furoate and Oxymetazoline.
  Interventions: Drug: mometasone furoate + Oxymetazoline

INTERVENTIONS:
Drug: mometasone furoate — 50μg, 1 puff in each nostril every evening
  Other Names: NASONEX
  Arms: mometasone furoate
Drug: Placebo — 1 puff in each nostril every evening
  Arms: Placebo
Drug: Oxymetazoline + Placebo — 1 puff of Oxymetazoline +1 puff of Placebo in each nostril every evening
  Other Names: Oxymetazoline Hydrochloride Spray + Placebo
  Arms: Oxymetazoline + Placebo
Drug: Placebo + placebo — 1 puff of placebo +1 puff of Placebo in each nostril every evening
  Other Names: Placebo
  Arms: Placebo + placebo
Drug: mometasone furoate + Placebo — 1 puff of mometasone furoate +1 puff of Placebo in each nostril every evening
  Other Names: NASONEX + Placebo
  Arms: mometasone furoate + Placebo
Drug: mometasone furoate + Oxymetazoline — 1 puff of mometasone furoate +1 puff of Oxymetazoline in each nostril every evening
  Other Names: NASONEX + Oxymetazoline Hydrochloride Spray
  Arms: mometasone furoate + Oxymetazoline

SUMMARY:
The purpose of this study is to determine the effect of MF/OXY in the treatment of adenoid hypertrophy children with severe allergic rhinitis.

DETAILED DESCRIPTION:
The investigators performed a two stages, parallel, randomized, double-blind, double-dummy, clinical trial in 240 AH children concomitant with perennial allergic rhinitis. In the first treatment stage, the 240 children were assigned to MF (50μg, 1 puff in each nostril every evening) or control group (normal saline) after two week's run-in period. After 6 week's treatment, the children in MF group were evaluated and grouped as responders and non-responders according to subjective symptoms and objective performance.

Responders were followed up for six months and reassessed. Non-responders underwent 2-week washout period and were randomly assigned to 4 groups receiving the following treatments: placebo, OXY (0.05%, 1 puff in each nostril every evening) or MF (50μg, 1 puff in each nostril every evening). All participants received 8 weeks' MF or its placebo plus one week's OXY or its placebo for every second week. After that, the patients were followed for six months and the evaluation was done at different time points.

ELIGIBILITY:
Inclusion Criteria:

* adenoid occluding at least 75% of the nasopharynx at nasal endoscopy
* age between 5 and 11 years
* chronic obstructive nasal symptoms no less than 12 months
* moderate-to-severe AR

Exclusion Criteria:

* tonsillar hypertrophy
* upper respiratory infection within the last 2 weeks
* sinonasal anatomic anomalies or diseases
* craniofacial malformations
* genetic diseases (i.e., Down's syndrome)
* neurologic or cardiovascular diseases
* immunodeficiency
* history of epistaxis
* asthma
* hypersensitivity to MF or OXY
* undergoing intranasal, topical, or systemic steroid or antibiotic treatment within the past 4 weeks

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
symptom score assessed by TNSS scopring system | six months

SECONDARY OUTCOMES:
adenoid size assessed by nasopharyngoscope （calculated the adenoid area in relation to the nasopharyngeal area） | six months
nasal volume assessd by Acoustic rhinometry | six months

CONTACTS AND LOCATIONS:
Overall Officials: renzhong Luo, Study Chair — Guangzhou Women and Children's Medical Center